CLINICAL TRIAL: NCT04320797
Title: Phenotype of Urinary CD4+ T Cells as Biomarkers for Prediction of Outcome in Lupus Nephritis
Brief Title: Urinary T Cell Biomarker for Prediction in Lupus Nephritis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Berlin Institute of Health (Other)
Responsible Party: Principal Investigator, Philipp Enghard, PD Dr. med., Charite University, Berlin, Germany
Other Study IDs: SLEFLURINOCYTE
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Lupus Nephritis
Keywords: lupus nephritis; systemic lupus erythematodes; urinary biomarker; outcome; prediction; urinary effector memory T lymphocytes; glomerulonephritis; non-invasive biomarker; flow cytometry; treatment outcome; CD4-positive T-lymphocytes/immunology
MeSH Terms: conditions — Lupus Nephritis; Glomerulonephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine, lymphocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active lupus nephritis: Patients with proliferative lupus nephritis (Class III and IV)
  Interventions: Diagnostic Test: Flow cytometry analysis of urine samples
- Control: Patients with systemic lupus erythematodes without lupus nephritis or lupus nephritis I, II or VI
  Interventions: Diagnostic Test: Flow cytometry analysis of urine samples

INTERVENTIONS:
Diagnostic Test: Flow cytometry analysis of urine samples — Urine samples will be conserved and frozen upon arrival. All samples will be stained according to T cell and TEC (tubular epithelial cells) panel with fluorochromes.
  T cell panel: CD3, CD4, CD8, CCR7, CD45RO, CD28, CD279; TEC panel: vimentin, cytokeratine, CD10, CD13, CD227, CD326

SUMMARY:
Urinary T-lymphocytes may be predictive for clinical outcome in patients with lupus nephritis. The investigators hypothesize that the amount of CD4+ effector/memory T-cells in urine at time of diagnosis predicts the outcome of patients with active lupus nephritis (LN) after 6 months of therapy. In a prospective, six-months follow-up study patients' urine will be analysed by flow cytometry every 60 days (+/- 10d). Treatment will be performed to the discretion of the treating clinician. After 6 months of treatment response will be determined as either complete response or partial response.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven lupus nephritis
* In absence of a biopsy a SLEDAI of at least 10 & at least two renal elements of the renal SLEDAI (rSLEDAI)
* Informed consent
* Diagnosis of SLE according to the American College of Rheumatology (ACR) criteria

Exclusion Criteria:

* Biopsy-proven non-SLE related disease
* Urinary tract infection
* Active menstrual bleeding
* Kidney transplantation during observation time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at medical wards of Charité Universitätsmedizin Berlin and University College London
Sampling Method: Probability Sample
Enrollment: 79 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Phenotype of CD4+ T cells at time point 0 predictive of clinical outcome in patients with lupus nephritis | 6 months
  Urinary CD4+ effector/memory T cell counts at time point 0 (time of diagnosis) predict clinical outcome (complete or partial response) after 6 months of treatment in patients with lupus nephritis. The frequency of effector/memory CD4+ T lymphocytes is higher in patients with non- or partial response.
  * Complete response at 24 weeks: the return to within 10 percent of normal values of serum creatinine levels, proteinuria, and urine sediment.
  * Partial response at 24 weeks: improvement of 50 percent in all abnormal renal measurements, without worsening - within 10 percent - of any measurement

SECONDARY OUTCOMES:
Distinction between proliferative LN (class III and class IV) and non-proliferative LN (classes I, II and VI) | 6 months
Analysis of patient with persistent renal abnormalities as partial response | 6 months
Prediction of complete or partial response according to normalization of the amount of urinary T cells at time point 2 and 4 | 6 months
Phenotype of CD8+ T cells at time point 0 predictive of clinical outcome in patients with lupus nephritis | 6 months
  Urinary CD8+ effector/memory T cell counts at time point 0 (time of diagnosis) predict clinical outcome (complete or partial response) after 6 months of treatment in patients with lupus nephritis. The frequency of effector/memory CD8+ T lymphocytes is higher in patients with non- or partial response.
Diagnosis of proliferative lupus nephritis in patients with systemic lupus erythematodes (SLE) | 6 months
  Diagnosis according to initial T cell count

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Enghard, PD Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Charité - Universitätsmedizin Berlin, Berlin, Germany
- The Royal Free London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Enghard P, Rieder C, Kopetschke K, Klocke JR, Undeutsch R, Biesen R, Dragun D, Gollasch M, Schneider U, Aupperle K, Humrich JY, Hiepe F, Backhaus M, Radbruch AH, Burmester GR, Riemekasten G. Urinary CD4 T cells identify SLE patients with proliferative lupus nephritis and can be used to monitor treatment response. Ann Rheum Dis. 2014 Jan;73(1):277-83. doi: 10.1136/annrheumdis-2012-202784. Epub 2013 Mar 8. PMID 23475982
- [Background] Arazi A, Rao DA, Berthier CC, Davidson A, Liu Y, Hoover PJ, Chicoine A, Eisenhaure TM, Jonsson AH, Li S, Lieb DJ, Zhang F, Slowikowski K, Browne EP, Noma A, Sutherby D, Steelman S, Smilek DE, Tosta P, Apruzzese W, Massarotti E, Dall'Era M, Park M, Kamen DL, Furie RA, Payan-Schober F, Pendergraft WF 3rd, McInnis EA, Buyon JP, Petri MA, Putterman C, Kalunian KC, Woodle ES, Lederer JA, Hildeman DA, Nusbaum C, Raychaudhuri S, Kretzler M, Anolik JH, Brenner MB, Wofsy D, Hacohen N, Diamond B; Accelerating Medicines Partnership in SLE network. The immune cell landscape in kidneys of patients with lupus nephritis. Nat Immunol. 2019 Jul;20(7):902-914. doi: 10.1038/s41590-019-0398-x. Epub 2019 Jun 17. PMID 31209404
- [Background] Dolff S, Abdulahad WH, Arends S, van Dijk MC, Limburg PC, Kallenberg CG, Bijl M. Urinary CD8+ T-cell counts discriminate between active and inactive lupus nephritis. Arthritis Res Ther. 2013 Feb 27;15(1):R36. doi: 10.1186/ar4189. PMID 23445537
- [Background] Kopetschke K, Klocke J, Griessbach AS, Humrich JY, Biesen R, Dragun D, Burmester GR, Enghard P, Riemekasten G. The cellular signature of urinary immune cells in Lupus nephritis: new insights into potential biomarkers. Arthritis Res Ther. 2015 Apr 3;17(1):94. doi: 10.1186/s13075-015-0600-y. PMID 25890061